CLINICAL TRIAL: NCT05974033
Title: IntraCranial Angiography-derived Fraction Flow-guided Percutaneous Transluminal Angioplasty and Stenting Versus Medical Therapy (ICAS-MT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICAS-MT
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: ICAS - Intracranial Atherosclerosis
Keywords: ICAS; Cerebral Arteriosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis | interventions — Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Stenting plus medical therapy
  Interventions: Combination Product: Stenting plus medical therapy
- Control group (Active Comparator): Medical therapy alone
  Interventions: Drug: Medical therapy alone

INTERVENTIONS:
Combination Product: Stenting plus medical therapy — Patients randomized to intervention group received the percutaneous transluminal balloon angioplasty with stenting within 5 days after randomization, and loading dose of aspirin and clopidogrel was allowed. Received aspirin, 100mg, plus clopidogrel, 75 mg, daily for 90 days after procedure.
  Arms: Intervention group
Drug: Medical therapy alone — Medical therapy alone: received aspirin, 100mg, plus clopidogrel, 75 mg, daily for 90 days after randomisation.
  Arms: Control group

SUMMARY:
A multicenter, open-label, blinded-endpoint, prospective, randomized controlled clinical trial with an "all comers" design.

DETAILED DESCRIPTION:
The main objective of this study is to investigate the impact of angiography-derived fractional flow (Angio-FF) on diagnostic and therapeutic decision-making in patients with symptomatic intracranial atherosclerotic stenosis (sICAS). The study aims to evaluate whether stenting plus medical therapy, compared to medical therapy alone, can benefit patients selected through Angio-FF screening.

For Group A, patients with significant stenosis and hemodynamic impairment identified through Angio-FF (≤0.7) screening are expected to have a higher risk. The patients will be enrolled in RCT trial, with a planned enrollment of 336 subjects.

For Group B, patients with significant stenosis but without hemodynamic impairment identified through Angio-FF (>0.7) screening will be included in the registry cohort, with a planned enrollment of 200 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥30 and ≤80 years old.
2. Symptomatic intracranial atherosclerotic stenosis: Transient ischemic attack (TIA) or stroke related to 70%-99% stenosis in the major intracranial arteries (intracranial segment of the internal carotid artery, M1 segment of the middle cerebral artery, V4 segment of the vertebral artery, and basilar artery) within the past 3 months.
3. Only one target vessel with 70-99% stenosis confirmed by angiography for enrollment in the trial (WASID criteria).
4. Patients with ischemic stroke should be performed with stenting beyond a duration of 2 weeks from the latest ischemic symptom onset, patients with TIA have no time restriction.
5. Pre-enrollment modified Rankin Scale (mRS) score ≤2.
6. Target vessel reference diameter must be measured to be 2 mm to 4.5 mm, target area of stenosis is less than or equal to 14mm in length.
7. Patients required to meet at least with one atherosclerotic risk factors, including hypertension, diabetes, hyperlipidemia, hyperhomocysteinemia, coronary heart disease, obesity, smoking history, and atherosclerosis in other arterial vessels.
8. Negative pregnancy test in a female who has had any menses in the last 18 months.
9. Patient is willing and able to return for all follow-up visits required by the protocol.
10. Patient understands the purpose and requirements of the study, can make him/herself understood, and has provided informed consent.

Exclusion Criteria:

1. Intracranial arterial stenosis not caused by atherosclerotic lesions, such as arterial dissection, moya-moya disease, vasculitic disease, viral vascular lesions (e.g., herpes zoster, varicella), neurosyphilis, other intracranial infections, radiation-induced vasculopathy, fibromuscular dysplasia, sickle cell disease, neurofibromatosis, benign central nervous system vascular diseases, postpartum angiopathy, suspected vasospastic process, suspected recanalized embolus, etc.
2. Any conditions that precludes proper angiographic assessment.
3. Preoperative MRI indicating only lacunar infarction in the target lesion territory.
4. History of subarachnoid hemorrhage, subdural or epidural hematoma within 30 days prior to enrollment, or untreated chronic subdural hematoma thickness≥5mm, or history of primary intracerebral hemorrhage.
5. At risk of hemorrhagic transformation during the procedure (CT or MRI showing infarct area diameter >5 cm); hemorrhagic transformation of an ischemic stroke within the past 15 days (detected by CT).
6. Tandem extracranial or intracranial stenosis (70%-99%) or occlusion that is proximal or distal to the target intracranial lesion
7. Bilateral intracranial vertebral artery stenosis of 70%-99% and uncertainty about which lesion is symptomatic (for example, if patient has pon, midbrain, temporal and occipital symptoms).
8. Stenting, angioplasty, or endarterectomy of an extracranial (carotid or vertebral artery) or intracranial artery within 30 days prior to expected enrollment date.
9. Previous treatment of target lesion with a stent, angioplasty, or other mechanical device, or plan to perform staged angioplasty followed by stenting of target lesion
10. Severe vascular tortuosity, severe calcification, or other factors that would preclude the safe introduction of a guiding catheter, guiding sheath or stent placement.
11. Presence of intraluminal thrombus proximal to or at the target lesion.
12. Any aneurysm proximal to or distal to intracranial stenotic artery.
13. Intracranial tumors or any intracranial vascular malformations.
14. Potential cardiac sources of emboli such as atrial fibrillation, left ventricular thrombus, heart valve replacement, atrial septal defect, ventricular septal defect, atrial myxoma, etc.
15. Myocardial infarction within previous 30 days.
16. Suspected severe allergy or contraindication to vascular interventional-related drugs or devices, such as aspirin, clopidogrel, general anesthesia agents, heparin, contrast agents, nitinol alloy, etc.
17. Active bleeding diathesis or coagulopathy, active gastrointestinal ulcer, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets count <100,000, hematocrit <30, INR >1.5, dysfunctions of the blood coagulation system.
18. uncontrolled severe hypertension (systolic BP>180mm Hg or diastolic BP>110mm Hg)
19. Severe comorbidities or unstable conditions, such as severe heart failure, respiratory failure, or renal failure (serum creatinine>264μmol/L, unless on dialysis), severe liver dysfunction (ALT or ALT >3 times normal), malignant tumors.
20. Major surgery performed within 30 days prior to enrollment or planned inpatient surgery within 90 days after enrollment.
21. Pregnancy or intent to become pregnant during the trial period.
22. Currently participating in another clinical trial.
23. Life expectancy less than 3 years
24. Patients unable to complete follow-up due to cognitive impairment, emotional disorders, or mental illness.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Stroke or death | Stroke or death within 30 days after enrollment; Or stroke in the territory of the symptomatic intracranial artery (SIT) between 30 days and 1 year.
  Stroke or death within 30 days after enrollment; Or stroke in the territory of the symptomatic intracranial artery (SIT) between 30 days and 1 year.

SECONDARY OUTCOMES:
Ischemic stroke in the target vessel territory | Within 1-3 years after enrollment
  Ischemic stroke in the target vessel territory
Ischemic stroke in non-target vessel territory | Within 30 days to 1 year, and within 1-3 years after enrollment
  Ischemic stroke in non-target vessel territory
Any occurrence of cerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage | Within 30 days to 3 years after enrollment
  Any occurrence of cerebral hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage
Any cause of death | Within 30 days to 3 years after enrollment
  Any cause of death
mRS score | At 1 year, 2 years, and 3 years after enrollment
  Modified Rankin scale (mRS) score. The value range 0-6: higher scores mean a worse outcome.
National Institutes of Health Stroke Scale (NIHSS) score | At 1 year, 2 years, and 3 years after enrollment
  Stroke severity (NIHSS score). The value range 0-42: higher scores mean a worse outcome.
Barthel Index | At 1 year, 2 years, and 3 years after enrollment
  An ordinal scale which measures a person's ability to complete activities of daily living. The value range 0-100: higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jianimin Liu, M.D., Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses
URL: http://www.ocin.org.cn/about